CLINICAL TRIAL: NCT02617771
Title: Impact of Vitamin D Supplementation on Recurrent Respiratory Infections in Paediatric
Brief Title: Impact of Vitamin D Supplementation on Recurrent Respiratory Infections in Paediatric Primary Care.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Prof. Maria Elisabetta Baldassarre, MD, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VITDBA1
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Recurrent Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vit D (Active Comparator): Vitamin D oral supplementation (400 UI/die up to 12 month or 600 UI/die beyond 1 year) from October to March
  Interventions: Drug: Vitamin D3
- Control (No Intervention)

INTERVENTIONS:
Drug: Vitamin D3 — from October to March, a Vitamin D oral supplementation (400 UI/die up to 12 month or 600 UI/die beyond 1 year
  Arms: Vit D

SUMMARY:
Up to date, some clinical trial have evaluated the efficacy and safety of Vitamin D supplementation in children with RRI, with no conclusive information.

Therefore, the investigators designed a prospective, single-blind, clinical trial to evaluate whether oral supplementation with vitamin D from October to April reduces the global health burden of recurrent respiratory tract infections in a primary care setting.

The primary outcome was evaluated if Vitamin D supplementation during autumn and winter can reduce the number of respiratory tract infections in children diagnosed with recurrent respiratory tract infections the seasons before.

Secondary objectives was the assessment of Vitamin D supplementation benefits on global socioeconomic burden of recurrent respiratory tract infections in a primary care setting, according to number of visits to the primary care paediatrician and use of antibiotics due to respiratory tract infections.

DETAILED DESCRIPTION:
The University study personnel randomly allocated patients to receive, from October to March, a Vitamin D oral supplementation (400 UI/die up to 12 month or 600 UI/die beyond 1 year) or not.

Randomization was performed using a free web-based service that offers random assignment; patients were randomized considering gender and age class (up to 12 months; beyond 1 years). The primary care practitioner was blinded regarding the study group allocation.

Inclusion criteria were: a) patients diagnosed the seasons before with: ≥ 6 respiratory infections per annum OR ≥ 1 respiratory infections per month involving the upper airways from September to April OR ≥ 3 respiratory infections per annum involving the lower airways. b) patients with no findings suggestive of an immunodeficiency on history and physical examination.

From the recruitment, parents recorded number and type of diagnosed respiratory tract infections, number of ambulatory visits, use of antibiotics and duration of symptoms in a structured diary.

Upper Respiratory Tract Infections (URTIs) comprehends diagnosis of acute otitis media, acute rhinosinusitis and acute pharyngotonsillitis. Lower Respiratory Tract Infections (LRTIs) comprehend diagnosis of bronchiolitis and pneumonia.

All parents had a close telephone contact to help them in the diary compilation. Adverse events related to the protocol were monitored. Missing data were recovered through the information system of the primary care practitioner.

Quantitative data were expressed as mean and standard deviation. To compare the mean between the two groups, Student's t-test for unpaired was used. The frequency of each visits to the pediatricians and use of antibiotics in the two group was calculated and expressed as a percentage. The χ² test was used to compare the percentages between the two groups. For all tests, P-values <0.05 were considered significant.

Since Italian National Health System covers all costs for pediatrician visits and antibiotics, cost assessment was made analysing the costs regarding the frequency of each parameters in treated and nontreated group. We considered as direct cost National Health System: Medical examination (20,66 euros for each examination, as provided by the Italian Ministry of Health) and use of Antibiotics (the cost was as in the list of the National Drug Authority).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed the seasons before with: ≥ 6 respiratory infections per annum
* ≥ 1 respiratory infections per month involving the upper airways from September to April
* ≥ 3 respiratory infections per annum involving the lower airways

Exclusion Criteria:

* patients with findings suggestive of an immunodeficiency on history and physical examination

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of recurrent respiratory tract infections for each months of study | From October 1, 2014, and March 31, 2015, up to 6 months
  reduction of the number of respiratory tract infections in children diagnosed with recurrent respiratory tract infections the seasons before

SECONDARY OUTCOMES:
Cost assessment in euros according to antibiotics, paediatric visits and vitamin D supplementation | From October 1, 2014, and March 31, 2015, up to 6 months
  Secondary objectives was the assessment of Vitamin D supplementation benefits on global socioeconomic burden of recurrent respiratory tract infections in a primary care setting, according to number of visits to the primary care paediatrician and use of antibiotics due to respiratory tract infections.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisabetta Baldassarre, MD, Principal Investigator — University of Bari

REFERENCES:
- [Background] de Sa Del Fiol F, Barberato-Filho S, Lopes LC, de Cassia Bergamaschi C. Vitamin D and respiratory infections. J Infect Dev Ctries. 2015 Apr 15;9(4):355-61. doi: 10.3855/jidc.5711. PMID 25881523
- [Result] Zittermann A, Gummert JF. Nonclassical vitamin D action. Nutrients. 2010 Apr;2(4):408-25. doi: 10.3390/nu2040408. Epub 2010 Mar 25. PMID 22254030